CLINICAL TRIAL: NCT03602898
Title: A Randomized Phase II Study to Compare ATG or Post-Transplant Cyclophosphamide to Calcineurin Inhibitor-Methotrexate as GVHD Prophylaxis After Myeloablative Unrelated Donor Peripheral Blood Stem Cell Transplantation
Brief Title: Comparing ATG or Post-Transplant Cyclophosphamide to Calcineurin Inhibitor-Methotrexate as GVHD Prophylaxis After Myeloablative Unrelated Donor Peripheral Blood Stem Cell Transplantation
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient funding
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9954; NCI-2018-01302 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9954 (Other: Fred Hutch/University of Washington Cancer Consortium); RG1001747 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2018-07-13; First posted 2018-07-27 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Acute Lymphoblastic Leukemia in Remission; Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Chronic Myelomonocytic Leukemia; Chronic Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Hematopoietic and Lymphoid System Neoplasm; Myelodysplastic Syndrome; Myelofibrosis; Myeloproliferative Neoplasm; Recurrent Acute Myeloid Leukemia; Recurrent Hodgkin Lymphoma; Recurrent Non-Hodgkin Lymphoma; Refractory Acute Myeloid Leukemia; Therapy-Related Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Myelodysplastic Syndromes; Primary Myelofibrosis; Myeloproliferative Disorders; Leukemia, Myeloid, Acute; Hodgkin Disease; Lymphoma, Non-Hodgkin | interventions — Antilymphocyte Serum; Busulfan; Cyclophosphamide; Cyclosporine; Cyclosporins; fludarabine phosphate; Methotrexate; merphos; Peripheral Blood Stem Cell Transplantation; Tacrolimus; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1 (ATG, tacrolimus or cyclosporine, methotrexate) (Experimental): Participants receive conditioning regimen (see detailed description) and then undergo peripheral blood stem cell transplantation on day 0. Participants receive anti-thymocyte globulin IV over 4-6 hours on days -3 to -1. Beginning day -1, participants also receive tacrolimus IV or cyclosporine IV BID tapered at day 50, and methotrexate IV on days 1, 3, 6 and 11 in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Anti-Thymocyte Globulin; Drug: Busulfan; Drug: Cyclophosphamide; Drug: Cyclosporine; Drug: Fludarabine Phosphate; Drug: Methotrexate; Procedure: Peripheral Blood Stem Cell Transplantation; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Tacrolimus; Radiation: Total-Body Irradiation
- Arm 2 (cyclophosphamide, tacrolimus or cyclosporine) (Experimental): Participants receive conditioning regimen (see detailed description) and then undergo peripheral blood stem cell transplantation on day 0. Participants receive cyclophosphamide IV over 1-2 hours on days 3 and 4. Beginning day 5, participants also receive tacrolimus IV or cyclosporine IV BID tapered at day 50 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Busulfan; Drug: Cyclophosphamide; Drug: Cyclosporine; Drug: Fludarabine Phosphate; Procedure: Peripheral Blood Stem Cell Transplantation; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Tacrolimus; Radiation: Total-Body Irradiation
- Arm 3 (tacrolimus or cyclosporine, methotrexate) (Experimental): Participants receive conditioning regimen (see detailed description) and then undergo peripheral blood stem cell transplantation on day 0. Beginning day -1, participants receive tacrolimus IV or cyclosporine IV BID tapered at day 50, and methotrexate IV on days 1, 3, 6 and 11.
  Interventions: Drug: Busulfan; Drug: Cyclophosphamide; Drug: Cyclosporine; Drug: Fludarabine Phosphate; Drug: Methotrexate; Procedure: Peripheral Blood Stem Cell Transplantation; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Tacrolimus; Radiation: Total-Body Irradiation

INTERVENTIONS:
Biological: Anti-Thymocyte Globulin — Given IV
  Other Names: Antithymocyte Globulin; Antithymocyte Serum; ATG; ATS
  Arms: Arm 1 (ATG, tacrolimus or cyclosporine, methotrexate)
Drug: Busulfan — Given IV or PO
  Other Names: 1, 4-Bis[methanesulfonoxy]butane; BUS; Bussulfam; Busulfanum; Busulfex; Busulphan; CB 2041; CB-2041; Glyzophrol; GT 41; GT-41; Joacamine; Methanesulfonic Acid Tetramethylene Ester; Methanesulfonic acid, tetramethylene ester; Mielucin; Misulban; Misulfan; Mitosan; Myeleukon; Myeloleukon; Myelosan; Mylecytan; Myleran; Sulfabutin; Tetramethylene Bis(methanesulfonate); Tetramethylene bis[methanesulfonate]; WR-19508
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Cyclosporine — Given IV or PO
  Other Names: 27-400; Ciclosporin; CsA; Cyclosporin; Cyclosporin A; Gengraf; Neoral; OL 27-400; Sandimmune; SangCya
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Drug: Methotrexate — Given IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
  Arms: Arm 1 (ATG, tacrolimus or cyclosporine, methotrexate); Arm 3 (tacrolimus or cyclosporine, methotrexate)
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo peripheral blood stem cell transplantation
  Other Names: PBPC transplantation; PBSCT; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplant; Peripheral Stem Cell Transplantation
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Drug: Tacrolimus — Given IV or PO
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: Total Body Irradiation; whole body irradiation; Whole-Body Irradiation; TBI

SUMMARY:
This phase II trial studies how well 3 different drug combinations prevent graft versus host disease (GVHD) after donor stem cell transplant. Calcineurin inhibitors, such as cyclosporine and tacrolimus, may stop the activity of donor cells that can cause GVHD. Chemotherapy drugs, such as cyclophosphamide and methotrexate, may also stop the donor cells that can lead to GVHD while not affecting the cancer-fighting donor cells. Immunosuppressive therapy, such as anti-thymocyte globulin (ATG), is used to decrease the body's immune response and reduces the risk of GVHD. It is not yet known which combination of drugs: 1) ATG, methotrexate, and calcineurin inhibitor 2) cyclophosphamide and calcineurin inhibitor, or 3) methotrexate and calcineurin inhibitor may work best to prevent graft versus host disease and result in best overall outcome after donor stem cell transplant.

DETAILED DESCRIPTION:
OUTLINE:

CONDITIONING REGIMENS: Participants receive 1 of 3 regimens and are randomized to 1 of 3 arms for GVHD prophylaxis.

REGIMEN A: Participants undergo total body irradiation (TBI) twice daily (BID) on days -6 to -4 (-7 to -4 for those < 18 years), then receive cyclophosphamide IV over 1-2 hours on days -3 and -2. Participants randomized to Arm 2 only receive TBI on days -3 to -1 (-4 to -1 for those < 18 years).

REGIMEN B: Participants receive fludarabine phosphate IV and busulfan IV every 6 hours on days -5 to -2.

REGIMEN C: Participants receive busulfan orally (PO) or IV every 6 hours on days -7 to -4 and cyclophosphamide IV over 1-2 hours on days -3 and -2.

Myelofibrosis or other myeloproliferative neoplasms: Participants >= 18 years receive cyclophosphamide IV over 1-2 hours on days -7 and -6 and busulfan IV on days -5 to -2. Participants < 17 years receive busulfan IV every 6 hours on days -7 to -4 and cyclophosphamide IV on days -3 and -2.

All participants undergo peripheral blood stem cell transplantation on day 0.

ARM 1: Participants receive anti-thymocyte globulin IV over 4-6 hours on days -3 to -1. Beginning day -1, participants also receive tacrolimus IV or cyclosporine IV twice daily (BID) tapered at day 50, and methotrexate IV on days 1, 3, 6 and 11 in the absence of disease progression or unacceptable toxicity.

ARM 2: Participants receive cyclophosphamide IV over 1-2 hours on days 3 and 4. Beginning day 5, participants also receive tacrolimus IV or cyclosporine IV BID tapered at day 50 in the absence of disease progression or unacceptable toxicity.

ARM 3: Beginning day -1, participants receive tacrolimus IV or cyclosporine IV BID tapered at day 50, and methotrexate IV on days 1, 3, 6 and 11 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up at 6 months, then annually up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* The following diseases will be permitted, although other diagnoses can be considered if approved by Fred Hutch Patient Care Conference or the participating institution's patient review committees and the principal investigator:

  * Acute lymphocytic leukemia (ALL) in complete remission (CR)1 with high risk features defined as evidence of adverse cytogenetics such as t(9;22), t(1;19), t(4;11), or MLL rearrangements or presence of minimal residual disease
  * Acute myeloid leukemia (AML) in CR1 with high risk features defined as:

    * Intermediate or adverse risk disease as defined by European LeukemiaNet (ELN) 2017
    * Greater than 1 cycle of induction therapy required to achieve remission
    * Preceding myelodysplastic syndrome (MDS) or myelofibrosis
    * Therapy-related AML
    * Presence of FLT3 internal tandem duplications
    * French-American-British (FAB) M6 or M7 classification
  * Acute leukemia (ALL or AML) in second (2nd) or greater CR (CR ≥ 2)
  * Refractory or relapsed AML with =< 5% bone marrow blasts and no circulating blasts by morphology or proven extramedullary disease
  * Myelodysplastic syndrome (MDS) with following high risk features: poor cytogenetics (-7, inv(3)/t(3q)/del(3q), del(7q) or complex cytogenetics defined as >= 3 abnormalities), Revised International Prognostic Scoring System (IPSS-R) risk group intermediate or higher, or treatment-related MDS
  * Any phase of MDS if patient is < 21 years of age
  * Chronic myelogenous leukemia (CML) beyond 1st chronic phase or resistant to tyrosine kinase inhibitors (adults)
  * Chronic myelomonocytic leukemia (CMML)
  * Myeloproliferative disorders/myelofibrosis
  * Hodgkin or non-Hodgkin lymphoma: relapsed chemotherapy-sensitive (complete or partial response)
* Female patients must have negative standard pregnancy test (all women of child bearing-potential must have test performed)
* Ability to understand and the willingness to sign a written informed consent document
* For patients with acute leukemia, CR is defined as =< 5% marrow blasts by morphology. CR with incomplete count recovery is allowed
* DONOR INCLUSION
* Unrelated donors matched for human leukocyte antigen (HLA)-A, B, C, DRB1 and DQB1 by high resolution typing
* Donors are excluded when preexisting immunoreactivity is identified that would jeopardize donor hematopoietic cell engraftment. This determination is based on the standard practice of the individual institution. The recommended procedure for patients with 10 of 10 HLA allele level (phenotypic) match is to obtain a panel reactive antibody (PRA) screens to class I and class II antigens for all patients before hematopoietic cell transplantation (HCT). If the PRA shows > 10% activity, then flow cytometric or B and T cell cytotoxic cross matches should be obtained. The donor should be excluded if any of the cytotoxic cross match assays are positive
* Only granulocyte colony-stimulating factor (G-CSF) mobilized peripheral blood stem cell (PBSC) will be permitted as a hematopoietic stem cell (HSC) source on this protocol
* Donors must meet the selection criteria for administration of G-CSF and apheresis defined based on each institution's standard practice protocol for unrelated donors
* Donors must be capable of giving informed consent

Exclusion Criteria:

* Prior autologous or allogeneic stem cell transplant
* Performance status: Karnofsky score <60 or Lansky score <50 for patients <16 years old
* Uncontrolled infection. The protocol principal investigator (PI) will be final arbiter if there is uncertainty regarding whether a previous infection is under adequate control to allow enrollment in the study
* Positive serology for human immunodeficiency virus (HIV)-1, 2 or human T-lymphotropic virus (HTLV)-1, 2
* Left ventricular ejection fraction < 45%. Uncontrolled arrhythmias or symptomatic cardiac disease
* Symptomatic pulmonary disease. Forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC), diffusion capacity of the lung for carbon monoxide (DLCO) =< 50% of predicted (corrected for hemoglobin). Use of continuous supplemental oxygen
* Calculated (Cockroft-Gault; or appropriate calculation for pediatric patients) serum creatinine clearance <60 mL/min. If the calculated CrCl is 50-60 mL/min, but a measured CrCl by 24 hour urine collection is > 60 mL/min, this measurement is acceptable
* Total serum bilirubin more than twice upper normal limit
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) more than 3-fold higher than laboratory upper normal limits
* History of allergy or anaphylactic reaction to rabbit protein or to any product excipients
* Subjects may not be enrolled in other investigational trials with acute or chronic GVHD as the primary endpoint
* DONOR EXCLUSION
* Donor who will exclusively donate marrow
* Donors who are HIV-positive
* Potential donors who for psychological, physiological, or medical reasons cannot tolerate administration of G-CSF or apheresis
* Donors who are allergic to filgrastim or Escherichia (E.) coli-derived proteins
* Donor-related risks to recipients
* Positive anti-donor lymphocytotoxic crossmatch
* Pregnant or lactating women
* Prior malignancy within the last 5 years

Max Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2023-09-17 (Estimated); Study Completion 2023-09-17 (Estimated)

PRIMARY OUTCOMES:
Moderate to severe chronic graft versus host disease (GVHD) based on National Institute of Health 2014 consensus criteria | At 1 year
  Probabilities of chronic GVHD at one year will be compared using a chi-square test.

SECONDARY OUTCOMES:
Survival | At 1 year post transplant
GVHD-free relapse-free survival (GRFS) | At 1 year post transplant
Chronic GVHD-free relapse-free survival (CRFS) | At 1 year post transplant
Grade II-IV acute GVHD | At 100 days
Grade III-IV acute GVHD | At 100 days
Relapse | At 1 year post transplant
Non-relapse mortality | At 1 year post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Masumi Ueda Oshima, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No